CLINICAL TRIAL: NCT06117631
Title: First Thousand Days: Prevention of Early Life Obesity in Latino Infants and Toddlers
Brief Title: Project Sueño: Sleep & Understanding Early Nutrition in Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Megan Gray, Associate Professor of Pediatrics and Population Health, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00003961
Record Dates: First submitted 2023-05-09; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Infant Overweight; Infant Obesity; Infant Overnutrition; Infant Development; Metabolic Syndrome; Diabetes Mellitus Risk
Keywords: infant feeding; infant sleep; parenting practices; rapid weight gain; intergenerational obesity; diabetes prevention
MeSH Terms: conditions — Pediatric Obesity; Infant Nutrition Disorders; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Centering Parenting (Experimental): At each well-child check from 2- to 24-months, a trained bilingual facilitator from the CommUnityCare Centering Parenting program will present curriculum in person during 2-hour visits in a room with 3-8 mother-baby pairs per group. During each session, each mother-baby pair will be pulled out to a private medical room for a brief individual well child appointment with the pediatrician. During this appointment, infant measurements, physical exam, and discussion of unique concerns will take place before the pair returns to the session. There are 8 scheduled well child checks by the age of two, where regular parenting topics will be covered (i.e. discipline, safety, co-parenting, sibling relationships, childcare, development). Each Centering session is expected to last approximately 2 hours, for a total commitment of approximately 16 hours across 8 group sessions over the course of 22 months for each participant. Total time of enrollment should be approximately 22-24 months.
  Interventions: Behavioral: Centering Parenting
- Group B: Bright by Text (Active Comparator): This group will receive standard of care individual well child checks with their regular CommUnityCare pediatrician, with standard anticipatory guidance on feeding and sleep. Additionally, this group will be enrolled in a text-based parenting coaching program. The Bright by Text program will provide parenting tips two to three times weekly; tailored through community partner United Way of Central Texas offering local parent support and resources. The Bright by Text program is a message subscription program rather than an application. Participants may decide on their own how much to engage with the text-based program, so total time commitment cannot be estimated. Total time of enrollment should be approximately 22-24 months.
  Interventions: Behavioral: Bright by Text
- Group C: Standard of Care (No Intervention): This group will receive standard of care individual well child checks with their regular pediatrician, with standard anticipatory guidance on feeding and sleep. Total time of enrollment should be approximately 22-24 months.

INTERVENTIONS:
Behavioral: Centering Parenting — See Arm description.
  Arms: Group A: Centering Parenting
Behavioral: Bright by Text — See Arm description.
  Arms: Group B: Bright by Text

SUMMARY:
The purpose of the study is to understand how mothers think and feel about feeding their babies and putting them to sleep, understand more about programs that can support mothers taking care of babies, and how professionals can be most helpful in helping mothers make decisions about their baby's feeding and sleeping. The overarching goal is to prevent early life obesity and progression to metabolic syndrome in high-risk populations, starting with healthy toddler weights by age 2 years.

DETAILED DESCRIPTION:
This study seeks to intervene just in time for families at highest risk of early life obesity and obesity-related comorbidities (such as Type 2 diabetes), to prevent intergenerational obesity and metabolic syndrome for Hispanic families. For those children exposed to gestational diabetes (GDM) or maternal overweight/obesity in utero, there is a critical need for effective early life strategies for secondary prevention of obesity, to interrupt intergenerational transmission. This study will offer community-embedded coaching to families learn how to responsively feed their babies using 2 models: group visits and text-based. The investigators will also assess responsive sleep practices; i.e. paying attention to an infant's sleep cues as well as hunger cues, breaking the feeding to sleep association, and not overfeeding at night. Infant and toddler sleep, both duration and quality, has not been well studied in this population for early life obesity prevention. This study is specifically exploring pathways from prenatal gestational diabetes and maternal overweight/obesity to dysregulated infant feeding and sleep. Few interventions around infant sleep exist for the Hispanic population, or resources in Spanish-language around sleep coaching; let alone analyses on parents' self-efficacy and behavior change. In this study, the investigators aim to better understand the complex socioenvironmental drivers of infant sleep and feeding behaviors, and the prenatal risks related to infant rapid weight gain, in order to target modifiable factors in this population.

ELIGIBILITY:
Inclusion Criteria:

* Mother to infant born full term > 37 weeks, and are under 1 month of age
* Infant is singleton
* Infant has no identified health problems
* Infant is patient of CommUnityCare
* Mother is 18 years of age
* Mother is Latino/Hispanic ethnicity
* Mother is willing to commit to study follow-up visits

Exclusion Criteria:

* Mother smokes
* Mother works primarily at night
* Infant has metabolic or chromosomal disorders, chronic neurological or respiratory conditions, or developmental disability

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess impact of group-based parent support coaching on infant feeding practices in first 2 years of child's life. | 2- to 24-months of infant age
  Assessment instruments include: Complementary Feeding History questionnaire, Nutrition Data System for Research, Expanded Food and Nutrition Education questionnaire, Infant Feeding Style Questionnaire.
Assess impact of text-based parent support coaching on infant feeding practices in first 2 years of child's life. | 2- to 24-months of infant age
  Assessment instruments include: Complementary Feeding History questionnaire, Nutrition Data System for Research, Expanded Food and Nutrition Education questionnaire, Infant Feeding Style Questionnaire.
Assess impact of group-based parent support coaching in first 2 years of child's life on responsive feeding and healthy sleep practices. | 2- to 24-months of infant age
  Assessment of parental responsive feeding practices, and infant sleep and temperament. Assessment instruments include: Complementary Feeding History questionnaire, Nutrition Data System for Research, Expanded Food and Nutrition Education questionnaire, Infant Feeding Style Questionnaire, Brief Infant Sleep Questionnaire, Children's Sleep Habits Questionnaire, Infant Toddler Temperament Tool. Sleep will additionally be assessed using 1-week sleep diaries and accelerometry at 2-, 6-, 12-, 18-, and 24-months of age.
Assess impact of text-based parent support coaching in first 2 years of child's life on responsive feeding and healthy sleep practices. | 2- to 24-months of infant age
  Assessment of parental responsive feeding practices, and infant sleep and temperament. Assessment instruments include: Complementary Feeding History questionnaire, Nutrition Data System for Research, Expanded Food and Nutrition Education questionnaire, Infant Feeding Style Questionnaire, Brief Infant Sleep Questionnaire, Children's Sleep Habits Questionnaire, Infant Toddler Temperament Tool. Sleep will additionally be assessed using 1-week sleep diaries and accelerometry at 2-, 6-, 12-, 18-, and 24-months of age.
Determine how parent support coaching and other predictors relate to infant and toddler growth in Latino children in first 2 years of life. | 2- to 24-months of infant age
  Assessment of variability of growth patterns by modeling of trajectories of weight gain in first 2 years of life.

CONTACTS AND LOCATIONS:
Overall Officials: Megan J Gray, MD,MPH,FAAP, Principal Investigator — University of Texas at Austin - Dell Medical School
Locations (1):
- CommUnity Care: North Central Health Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with individuals who are collaborating with the research team on this study; these investigators will be added to the IRB and/or only provided with a limited deidentified dataset.
  Limited, de-identified aggregate data will also be shared with the following data repositories:
  * National Sleep Research Resource (NSRR): will share physiological signals and de-identified clinical data
  * National Children's Study (NCS) Archive: will share intervention protocol and program feedback to serve as a guide for future interventions
  * Harvard Dataverse: will share qualitative data
Supporting Information: Study Protocol

REFERENCES:
- [Background] Lavner JA, Stansfield BK, Beach SRH, Brody GH, Birch LL. Sleep SAAF: a responsive parenting intervention to prevent excessive weight gain and obesity among African American infants. BMC Pediatr. 2019 Jul 5;19(1):224. doi: 10.1186/s12887-019-1583-7. PMID 31277694
- [Background] Baxter KA, Nambiar S, So THJ, Gallegos D, Byrne R. Parental Feeding Practices in Families Experiencing Food Insecurity: A Scoping Review. Int J Environ Res Public Health. 2022 May 5;19(9):5604. doi: 10.3390/ijerph19095604. PMID 35564998
- [Background] Gross RS, Mendelsohn AL, Arana MM, Messito MJ. Food Insecurity During Pregnancy and Breastfeeding by Low-Income Hispanic Mothers. Pediatrics. 2019 Jun;143(6):e20184113. doi: 10.1542/peds.2018-4113. Epub 2019 May 14. PMID 31088893
- [Background] Hall WA, Liva S, Moynihan M, Saunders R. A comparison of actigraphy and sleep diaries for infants' sleep behavior. Front Psychiatry. 2015 Feb 12;6:19. doi: 10.3389/fpsyt.2015.00019. eCollection 2015. PMID 25729371
- [Background] Van Hoorn M, Feuling MB, Allen K, Berry R, Brown S, Sullivan CM, Goday PS. Evaluation and Management of Reduced Dietary Diversity in Children with Pediatric Feeding Disorder. J Autism Dev Disord. 2023 Mar;53(3):1290-1297. doi: 10.1007/s10803-022-05715-8. Epub 2022 Aug 22. PMID 35996036
- [Background] Li X, Haneuse S, Rueschman M, Kaplan ER, Yu X, Davison KK, Redline S, Taveras EM. Longitudinal association of actigraphy-assessed sleep with physical growth in the first 6 months of life. Sleep. 2022 Jan 11;45(1):zsab243. doi: 10.1093/sleep/zsab243. PMID 34676870
- [Background] Yalcin SS, Tezol O, Caylan N, Erat Nergiz M, Yildiz D, Cicek S, Oflu A. Evaluation of problematic screen exposure in pre-schoolers using a unique tool called "seven-in-seven screen exposure questionnaire": cross-sectional study. BMC Pediatr. 2021 Oct 25;21(1):472. doi: 10.1186/s12887-021-02939-y. PMID 34696746
- [Background] Nadeau KJ, Anderson BJ, Berg EG, Chiang JL, Chou H, Copeland KC, Hannon TS, Huang TT, Lynch JL, Powell J, Sellers E, Tamborlane WV, Zeitler P. Youth-Onset Type 2 Diabetes Consensus Report: Current Status, Challenges, and Priorities. Diabetes Care. 2016 Sep;39(9):1635-42. doi: 10.2337/dc16-1066. Epub 2016 Aug 2. PMID 27486237

DOCUMENTS (1):
  • Informed Consent Form (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT06117631/ICF_000.pdf